CLINICAL TRIAL: NCT03613805
Title: Eversense and Dexcom G5 Comparison in Real Life: a Randomized Crossover Trial in Type 1 Diabetic Patients to Evaluate Differences in Accuracy, Efficacy and Quality of Life
Brief Title: Eversense and Dexcom G5: Efficacy and Accuracy in Type 1 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Daniela Bruttomesso, principal investigator, MD, PhD, Metabolic Unit, University of Padua, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 4270/AO/17
Record Dates: First submitted 2018-04-26; First posted 2018-08-03 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexcom G5 - Eversense (Active Comparator): Patients will wear first Dexcom G5 (Dexcom San Diego, CA, USA) transcutaneous sensor for 3 months, then Eversnese(Senseonics Inc, MD, USA) implantable sensor for 3 months Accuracy and efficacy will be evaluated
  Interventions: Device: Dexcom G5-Eversense
- Eversense- Dexcom G5 (Experimental): Patients will wear first Eversense (Senseonics Inc, MD, USA) implantable sensor for 3 months, then Dexcom G5 (Dexcom San Diego, CA, USA) transcutaneous sensor for 3 months accuracy and efficacy will be evaluated
  Interventions: Device: Eversense-Dexcom G5

INTERVENTIONS:
Device: Dexcom G5-Eversense — Patients will wear sensor for 3 months, monitor blood capillary values 4 times/day. At the beginning and at the end of the period HbA1c will be measured and questionnaires will be administered
  Arms: Dexcom G5 - Eversense
Device: Eversense-Dexcom G5 — Patients will wear sensor for 3 months, monitor blood capillary values 4 times/day. At the beginning and at the end of the period HbA1c will be measured and questionnaires will be administered.
  After 30-50 days of sensor implantation patients will wear also Dexcom G5 for a week to compare accuracy simultaneously
  Arms: Eversense- Dexcom G5

SUMMARY:
Continuous Glucose Monitoring (CGM) systems improve glycaemic control in type 1 diabetic patients but they have different characteristics that could influence patients' quality of life and glycaemic control.

In this randomized cross over study investigators will compare 2 different CGM systems: Eversense implantable sensor (Senseonics, Germantown, MD, USA) and the standard transcutaneous sensor Dexcom G5 (Dexcom, San Diego, CA, USA). Investigators will evaluate sensors' accuracy, impact on quality of life and efficacy in optimizing glycaemic control.

The investigator's study's results might help clinicians choose the sensor and evaluate how sensor differences could impact glycaemic control.

DETAILED DESCRIPTION:
Good glycaemic control in type 1 diabetic patients prevents the onset and progression of chronic complications. Continuous Glucose Monitoring (CGM) systems help patients improve glycaemic control by providing real-time glucose levels, glycaemic tendency, glycaemic swing rate and by alerting the patient when the glucose value read by the sensor reaches a predefined threshold of hyper or hypoglycaemia.

Several CGM systems are available and they have different characteristics that could influence patients' quality of life and glycaemic control.

In this randomized cross over study investigators will compare 2 different CGM systems: Eversense implantable sensor (Senseonics, Germantown, MD, USA) and the standard transcutaneous sensor Dexcom G5 (Dexcom, San Diego, CA, USA). Investigators will evaluate sensors' accuracy, impact on quality of life and efficacy in optimizing glycaemic control.

Patients will use Dexcom G5 or Eversense for three months, respectively, in a randomized order. Accuracy will be evaluated comparing sensors values with capillary blood glucose at home.

Quality of life will be assessed at the beginning and at the end of each three-month period through validated questionnaires to underline differences in different sensors use.

Time spent in target (70-180 mg/dl), in hypoglycamiea and hyperglycemia will be evaluated with both sensors to assess differences in glycaemic control induced by different alarm system and by the presence of predictive alarms

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of at least 18 years of age
* Diagnosis of type 1 diabetes mellitus (diagnosed according to World Health Organization criteria) for at least 1 year
* Body Mass Index (BMI) <35 kg / m²
* Availability to wear study equipment and to comply with the study protocol for its entire duration
* HbA1c <10%
* Signature of informed consent before any procedure related to the study.

Exclusion Criteria:

* Pregnancy, breastfeeding, intention to undergo pregnancy or refusal to use contraceptive methods during the study period (for female subjects).
* Known allergies to skin patches or disinfectants used during the study.
* Skin lesions, irritation, redness, edema in sites where sensors can be applied, as this might interfere with sensor's placement or with the accuracy of the glycaemic value detection.
* Use of drugs that may interfere with glucose metabolism (such as steroids) unless they are chronic therapies whose dosage has remained stable over the past 3 months and is expected to remain stable during the study period.
* Use of acetaminophen or other drugs that could influence sensor accuracy
* Severe medical or psychological conditions, which, in the opinion of the medical team, may compromise patients' safety while participating in the study.
* Patients enrolled in other clinical trials.
* Known disorders of adrenal glands, pancreatic tumors or insulinoma
* Patient's inability to comply with the procedures of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
device accuracy | after 3 months, at the end of the study for each arm of the study
  sensors' accuracy expressed in terms of MARD (mean absolute relative difference) versus capillary blood glucose in different glycaemic ranges

SECONDARY OUTCOMES:
Time spent in target | after 3 months, at the end of the study for each arm of the study
  % Time spent in target (70-180 mg/dl) using each sensor to evaluate sensor efficacy
HbA1c | after 3 months, at the end of the study for each arm of the study
  HbA1c changes using different sensors, to evaluate sensor efficacy
failure | after 3 months, at the end of the study for each arm of the study
  % Sensors' failure rate to evaluate sensor duration
Adverse events | after 3 months, at the end of the study for each arm of the study
  Adverse events (skin reactions, haematomas)
changes in quality of life | after 3 months, at the end of the study for each arm of the study
  DTSQ questionnaire
changes in fear of hypoglycaemia | after 3 months, at the end of the study for each arm of the study
  HFSII questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Italy